CLINICAL TRIAL: NCT02278601
Title: Comparison of Modified Programmed Intermittent Bolus (MPIB), Computer-integrated Patient Controlled Epidural Analgesia (CIPCEA) and Conventional Patient Controlled Epidural Analgesia (PCEA) During Labour
Brief Title: Comparison of Regimens MPIB, CIPCEA, PCEA
Acronym: COLEUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTGL13feb013
Record Dates: First submitted 2014-10-26; First posted 2014-10-30 (Estimated); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Breakthrough Pain
Keywords: Breakthrough pain
MeSH Terms: conditions — Breakthrough Pain | interventions — Ropivacaine; Fentanyl; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MPIB modified programmed intermittent bolus (Experimental): Modified programmed intermittent bolus (MPIB) up-down frequency of 5mls ropivacaine/fentanyl solution in bolus with epidural delivery system
  Interventions: Device: epidural delivery system; Drug: Ropivacaine; Drug: Fentanyl
- CIPCEA (Experimental): computer integrated patient controlled epidural analgesia (CIPCEA) up-down variable basal infusion of ropivacaine/fentanyl solution with epidural delivery system
  Interventions: Device: epidural delivery system; Drug: Ropivacaine; Drug: Fentanyl
- patient controlled epidural analgesia with basal infusion (Active Comparator): patient controlled epidural analgesia (PCEA) with fixed basal infusion of ropivacaine/fentanyl solution with epidural delivery system
  Interventions: Device: epidural delivery system; Drug: Ropivacaine; Drug: Fentanyl

INTERVENTIONS:
Device: epidural delivery system — epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution
Drug: Ropivacaine — epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution
  Other Names: amide local anaesthetic
Drug: Fentanyl — epidural delivery system for maintenance of labour epidural analgesia using 0.1% ropivacaine (amide local anaesthetic) with 2mcg/ml fentanyl (opioid) as maintenance solution
  Other Names: opioid

SUMMARY:
Epidural analgesia is the gold standard of pain relief for labour pain. Despite this, more than 50% of parturients continue to experience pain leading to suffering and increased caregiver workload. Women who have increased pain tend to have lower successful patient bolus demands when patient controlled epidural analgesia (PCEA) is utilised and have dysfunctional labour requiring obstetric intervention such as Caesarean or instrumental delivery. Labour pain often escalates and worsens as labour progresses requiring an individualized, variable, flexible analgesic regimen. Bolus epidural administrations have been shown to improve uniform spread of local anaesthetics with better pain relief, compared to fixed background infusions.

DETAILED DESCRIPTION:
The research team developed two novel epidural delivery regimens: computer-integrated PCEA (CIPCEA) and modified programmed intermittent bolus (MPIB) focused on individualization of analgesic requirements. This phase 3 double-blinded randomized controlled trial will compare the two novel regimens, and each with conventional PCEA with basal infusion (BI), in reducing breakthrough pain (failure of the regimen to provide adequate pain relief, necessitating unscheduled epidural supplementation) incidence as the primary outcome in nulliparous term women requesting labour epidural analgesia. In addition, a discrete choice experiment (DCE) in the format of a survey will be administered to estimate the women's preferences in treatment attributes related to epidural analgesia, including control over epidural dosage, chance of having breakthrough pain, motor block, instrumental delivery and out-of-pocket cost for epidural analgesia. We will also look into the association model for breakthrough pain that would take into account pre-delivery factors to better understand the mechanism of breakthrough pain during labor process.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (ASA physical status 1 and 2) nulliparous parturients at term (≥36 weeks gestation);
2. Singleton foetus
3. Early labour (cervical dilation ≤5cm)
4. Request labour epidural analgesia
5. At least 21 years of age

Exclusion Criteria:

1. parturients with multiple pregnancies
2. non-cephalic foetal presentation
3. obstetric (e.g. pre-eclampsia, premature rupture of amniotic membranes, gestational diabetes on insulin) and uncontrolled medical (e.g. cardiac disease) complications
4. have contraindications to neuraxial blockade or have received parenteral opioids with the last 2 hours.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 839 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Breakthrough pain | 1 day
  Unscheduled epidural supplementation by anaesthetist due to pain

SECONDARY OUTCOMES:
Number of subjects with Caesarean section | 1 day
  Number of subjects with Caesarean section
Number of subjects with Instrumental delivery | 1 day
  Number of subjects with Instrumental delivery (forceps, vacuum delivery)
Foetal outcome | 1 day
  APGAR scores
Willingness to pay | 1 day
  Discrete choice experiments (DCE) in survey format will be given to patients to determine patient's mean willingness to pay for epidural features, including control over epidural dosage, chance of having breakthrough pain, motor block, instrumental delivery and out-of-pocket cost for epidural analgesia)
Factors associated with epidural decisions | 1 day
  Participants will be exposed to 8 pairs of hypothetical medical scenarios as per the design of DCE. Participants have to choose the ideal scenario (A or B) that provides the highest perceived benefits. Each pair of scenarios represents a comprehensive combination of possible attributes related to epidural analgesia, including control over epidural dosage, chance of having breakthrough pain, motor block, instrumental delivery and out-of-pocket cost for epidural analgesia. The most common factors associated with optimal perceived benefits will be assessed based on these experimental design. A weighted estimate will be calculated for each attribute.
Pain vulnerability: Pain Catastrophizing Scale | 1 day
  Assessment will be done via Pain Catastrophizing Scale (PCS) questionnaire before delivery. Pain catastrophizing refers to the negative thought processes patients have when they are exposed to pain or painful experiences. The PCS is a 13-item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). It is broken into three subscales being magnification (0-12), rumination (0-16), and helplessness (0-24). A higher value in each subscale indicates a higher tendency to that subscale (worse outcome).
Edinburgh Postnatal Depression Scale before and after delivery | 5-9 weeks
  Assessment will be done via Edinburgh Postnatal Depression Scale (EPDS) before delivery, and again 5 to 9 weeks after delivery to assess patient's status on postnatal depression. The EPDS is a 10 item self-reported questionnaire validated for use as a screening tool for antenatal and postpartum depression in the clinical setting. Participants are asked to respond according to how they have felt in the past seven days, by which the questions correspond to common depressive symptoms. Each item is measured on a 4-point scale, with a total score in the range of 0 to 30. A higher total score indicates a greater degree of depressive symptoms. A score of 13 and above indicates clinically significant depressive symptom.
Sub-acute pain after childbirth | 5-9 weeks
  Assessment will be done via a pain survey at 5-9 weeks after delivery to ask on patient's pain experience, including the presence of sub-acute pain after childbirth, defined by presence or absence of pain that lasted for 4 weeks or more) (binary variable with categories "yes" or "no").

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Tan DJA, Lew JP, Jumhasan MB, Pang C, Sultana R, Sng BL. Investigating factors associated with success of breastfeeding in first-time mothers undergoing epidural analgesia: a prospective cohort study. Int Breastfeed J. 2018 Sep 5;13:42. doi: 10.1186/s13006-018-0184-7. eCollection 2018. PMID 30202425